CLINICAL TRIAL: NCT03077191
Title: Toxicity and Outcome of Whole Breast Hypofractionated Radiotherapy Without Boost: Results of a Homogeneous Single Institution Experience
Brief Title: Toxicity and Outcome of Whole Breast Hypofractionated Radiotherapy: a Single Institution Experience
Acronym: Ipomammella
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrei Fodor, MD, M.D., IRCCS San Raffaele
Other Study IDs: Ipomammella
Record Dates: First submitted 2017-02-16; First posted 2017-03-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Quality of Life; Radiotherapy; Adverse Effect, Dermatitis or Eczema; Survivorship
Keywords: hypofractionated whole breast radiotherapy; breast cancer; conservative treatment; quality of life
MeSH Terms: conditions — Breast Neoplasms; Dermatitis; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quality of life: Quality of life of breast cancer patients treated with conservative surgery (quadrantectomy) and adjuvant hypofractionated whole breast radiotherapy according to the institutional standard regimen, to a total dose of 40 Gy in 15 fraction over 3 weeks will be measured with EORTC quality of life questionnaires QLQ-C30 and QLQ-BR23, before the start of the radiotherapy, at the end of the radiotherapy and subsequently at every follow-up visit (the first at 6 months after the end of the treatment, then annually for 5 consecutive years after the first follow up visit).
  Interventions: Other: Quality of life measurement
- Breast cancer, retrospective: In the observational retrospective cohort patients with histologically confirmed breast cancer treated with hypofractionated/ultrahypofractionated radiotherapy to:
  * whole breast +/- Simultaneous Integrated Boost (SIB) to surgical bed,
  * breast/chest wall and lymph node areas +/- SIB to surgical bed,
  * surgical bed only, with accelerated partial breast irradiation,
  using 3D conformal radiotherapy or advanced radiotherapy techniques (IGRT, IMRT, SBRT) will be included.

INTERVENTIONS:
Other: Quality of life measurement — The quality of life of breast cancer patients treated with conservative surgery and adjuvant whole breast hypofractionated radiotherapy, without boost, will be evaluated.
  Groups: Quality of life

SUMMARY:
This is a homogeneous, single institution, observational, non-interventional, prospective study of 500 patients who will be treated according to the standard protocol of adjuvant hypofractionated radiotherapy after breast conserving surgery, at a total dose of 40 Gy/ 15 fr (5 fr/ week, 3 consecutive weeks). In addition to the regular follow up, the patients will respond to the quality-of-life questionnaires (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC), general, QLQ- C30, and specific for breast (BR), QLQ- BR23, at the first visit, at the end of radiotherapy and at the subsequent follow-up visits from 6 months up to 5 and a half years, to evaluate the quality of life during and after the treatment.

The study also has a retrospective arm of approximately 3300 patients (number of patients and characteristics of disease expanded with the amendment presented to the Lombardia 1 Ethics Committee in May 22/2024), treated from January 2009, for whom disease control and toxicity will be evaluated.

DETAILED DESCRIPTION:
The study is observational, homogeneous (performed in a single institution), non-interventional, and composed of two parts: one retrospective and one prospective (for which we request the registration in the register of clinical trials).

The patients with breast cancer treated with adjuvant hypofractionated radiotherapy at the Department of Radiotherapy of "San Raffaele Scientific Institute" (IRCCSSRaffaele) from January 2009 will be identified and their clinical and dosimetric data retrieved and analyzed.

The objectives of the retrospective arm of the study are the analysis, with a follow up of 5 years, of acute and late toxicity, and clinical outcomes, such as local and regional control, overall survival, disease free survival and cancer-specific survival. A secondary objective is the identification of prognostic factors for toxicity and disease progression.

With the amendment approved by the Ethics Committee 1 of Lombardy Region in 22/05/2024 (CET Em. 195-2024) the number of patients in the retrospective arm was expanded to 3300. Were included: patients treated with moderate hypofractionated or ultra-hypofractionated radiotherapy to whole breast+/- simultaneous integrated boost to surgical bed, patients treated with accelerated partial breast irradiation, patients treated with hypofractionated radiotherapy to regional nodal irradiation and whole breast+/-SIB to surgical bed. The follow-up period was expanded to 10 years.

The objective of the prospective arm of the study, for a cohort of 500 consecutive patients who agree to participate in the study, is to assess the quality of life of the patients treated with hypofractionated short course (3 weeks) radiotherapy. The quality-of-life questionnaires (QLQ) of the European organization for research and treatment of cancer (EORTC): QLQ-C30 (general) and QLQ-BR23 (specific for the breast), will be distributed before radiation treatment, at the time of patient enrollment, at the end of therapy and during the follow up visits, for a duration of 5 years after the first follow up, scheduled first at 6 months and then annually.

Given the non-interventional, observational nature of the study, the follow up program of the patients with breast cancer, treated according to the standard departmental protocol, will not be modified. The patients will be identified from the patient data base from medical records retrieved from the radiotherapy archive, and the images monitoring local evolution from the photo archive. The data will be extracted from medical records. In addition, the dosimetric data of the treatments will be recovered from the physical dosimetric archives and the extrapolated data will be correlated with clinical and toxicity outcomes.

For the patients of the prospective observational arm, the dosimetric data and quality of life questionnaires, as well as the follow up visit results, will be prospectively collected, registered in a data base, and subsequently analyzed.

The toxicity registered during the visits carried out during the treatment will be determined using the Radiation Therapy Oncology Group (RTOG) scale; the Scoring system of late effects of radiation on normal tissues (SOMA-LENT scale) will be used for toxicity registered during the follow up visits. The clinical points analyzed will include: quality of life, overall survival, disease free- and cancer specific-survival, local and regional control, distant metastasis free survival, acute and late toxicity, physical dosimetry and aesthetic results. The correlation between detected parameters will be evaluated for the identification of prognostic factors. Statistical analyses will be performed with SPSS software version 17.0 (SPSS Inc. Released 2008; SPSS Statistic for Windows, Version 17.0. Chicago, USA: SPSS Inc.) and MedCalc v.12.1.4.0 (MedCalc Software, Ostend, Belgium) and any updated version. Statistical tests to be used will include: uni- and multi-variate logistic regression to define predictors of incidence and prevalence of toxicity and local/ distant relapses; Cox model ( proportionally-hazard regression) uni- and multi-variate for actuarial analysis of predictors of toxicity and local/ distant relapses; Wilcoxon matched -pair test for the quality of life index variations; Spearman test for the correlation between continuous variables, ANOVA test for the effect of treatment variables on changes in QoL scores over time.

*Enrollment in the quality-of-life study was suspended in November 2021 due to patients' refusal to participate during the Sars-Cov2 pandemic, the adoption of shorter schedule protocols to minimize patient hospital visits, the adoption of a simultaneous integrated boost for patients with high risk of local relapse(TNBC, HER2+) requiring a change in the technique utilized.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with TNM Classification of Malignant Tumours pathological stage Tis-T4d, N0-N3, treated with surgery (conservative or mastectomy), accelerated partial breast irradiation or whole breast hypofractionated radiotherapy +/-SIB +/- regional lymph node irradiation

Exclusion Criteria:

- male breast cancer patients

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Study Population: Breast cancer patients treated with surgery (conservative/mastectomy), and hypofractionated/ultrahypofractionated radiotherapy to surgical bed or whole breast +/-SIB, +/- regional lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
quality of life after hypofractionated adjuvant radiotherapy | up to 66 months
  degree of general quality of life worsening of patients treated with hypofractionated adjuvant radiotherapy after breast conserving surgery assessed with EORTC quality of life questionnaires QLQ C30
breast specific quality of life after hypofractionated adjuvant radiotherapy | up to 66 months
  degree of specific quality of life worsening of patients treated with hypofractionated adjuvant radiotherapy after breast conserving surgery assessed with EORTC quality of life questionnaire QLQ BR23

SECONDARY OUTCOMES:
Local Relapse Free Survival | From the date of radiotherapy end until the date of local progression or date of death from any cause, whichever came first, assessed up to 120 months
  Local control of the disease (at the treated site)
Regional Relapse Free Survival | From the date of radiotherapy end until the date of regional progression or date of death from any cause, whichever came first, assessed up to 120 months
  Regional control (at the regional lymph node chains)
Distant Metastases Free Survival | From the date of radiotherapy end until the date of distant progression or date of death from any cause, whichever came first, assessed up to 120 months
  Distant metastasis developed after the treatment
Disease Free Survival | From the date of radiotherapy end until the date of first documented clinical progression or date of death from any cause, whichever came first, assessed up to 120 months
  Absence of disease progression during the follow-up
Cancer Specific Survival | From the date of radiotherapy end until the date of death from disease progression, assessed up to 120 months
  Cancer survival
Overall survival | From the date of radiotherapy end until the date death from any cause, assessed up to 120 months
  Survival from all causes
Acute toxicity | Up to three months from the start of radiotherapy
  Acute toxicity after hypofractionated whole breast adjuvant radiotherapy evaluated with CTCAE (Common Terminology Criteria for Adverse Events) scale v 5.0, which displayes grades from 1 to 5, with grade 1 mening mild toxicity and grade 5 death related to toxicity
Late toxicity | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 120 months
  Toxicity developed after three months until the end of follow-up or death, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity
Late skin toxicity | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 120 months
  Toxicity developed after three months until the end of follow-up or death, assessed with LENT-SOMA scale, which displayes grades from 1 to 4, with grade 1 meaning mild toxicity and grade 4 worst toxicity

OTHER OUTCOMES:
Aesthetic result | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 120 months
  Assessment of the effect of radiation therapy with photographs taken the day of treatment planning verification (before the first radiotherapy fraction), after 15 fractions of radiotherapy (at the end of radiation therapy), and during follow-up visits (the first 6 months after the end of radiotherapy and than at 18 months, 30 months, 42 months, 54 months and 66 months after the end of radiotherapy).
Predictive factor for disease progression and death | From radiotherapy end to date of local, regional progression, distant failure, or death, assessed up to 120 months
  actors predicting survival. Survival trees, univariate/multivariate Cox regression models will be estimated to identify potential risk factors associated with survival outcomes
Radiomic predictive factors for disease progression and death | From radiotherapy end to the first registered event (disease progression or death), assessed up to 120 months
  Simulation CT radiomic features predicting relapse or death will be extracted, acording to IBSI (Image Biomarker Standardisation Initiative), owning to the different families of features: Morphology, Statistical, Intensity Histogram, Grey Level Cooccurrence Matrix 3D-average, Grey Level Co-occurrence Matrix 3D-combined, Grey Level Run Lenght 3D-average. Grey Level Run Lenght 3D_combined, Grey Level Size Zone Matrix 3D, Neighbors Grey Tone Difference Matrix 3D, Grey Level Distance Zone Matrix 3D, standard convolutional filters within radiomic workflow (wavelets, Laplacian of Gaussian
Predictive factors for toxicity | From radiotherapy start until the end of follow-up or death, assessed up to 120 months
  Factors predicting toxicity. Survival trees, univariate/multivariate Cox regression models will be estimated to identify potential risk factors associated with toxicity
Radiomic predictive factors for toxicity | From radiotherapy start until the end of follow-up or death, assessed up to 120 months
  Simulation CT radiomic features predicting toxicity will be extracted, acording to IBSI (Image Biomarker Standardisation Initiative), owning to the different families of features: Morphology, Statistical, Intensity Histogram, Grey Level Cooccurrence Matrix 3D-average, Grey Level Co-occurrence Matrix 3D-combined, Grey Level Run Lenght 3D-average. Grey Level Run Lenght 3D_combined, Grey Level Size Zone Matrix 3D, Neighbors Grey Tone Difference Matrix 3D, Grey Level Distance Zone Matrix 3D, standard convolutional filters within radiomic workflow (wavelets, Laplacian of Gaussian)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Fodor, M.D., Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author (AF) will be evaluated by the Lombardy Territorial Ethics Committee 1.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for 2 years after the study closes
Access Criteria: Request from the corresponding author approved by the Lombardy Territorial Ethics Committee 1

REFERENCES:
- [Background] AIRTUM Working Group. I tumoti in Italia- Rapporto 2009. I trend dei tumori negli anni duemila ( 1998-2005). Epidemiol Prev 2009; 33(Suppl 1): 1-168.
- [Background] Ferlay J, Parkin DM, Steliarova-Foucher E. Estimates of cancer incidence and mortality in Europe in 2008. Eur J Cancer. 2010 Mar;46(4):765-81. doi: 10.1016/j.ejca.2009.12.014. Epub 2010 Jan 29. PMID 20116997
- [Background] http://www.istat.it/dati/dataset/20100129_00/
- [Background] Crocetti E; Airtum Working Group. [Numbers. Cancer survival in Italy is within the European average]. Epidemiol Prev. 2008 Jul-Oct;32(4-5):265. No abstract available. Italian. PMID 19186510
- [Background] Airtum Working Group. [Numbers (Airtum Working Group). Survival prospects change with time]. Epidemiol Prev. 2008 May-Jun;32(3):136. No abstract available. Italian. PMID 18828550
- [Background] Gotzsche PC, Nielsen M. Screening for breast cancer with mammography. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD001877. doi: 10.1002/14651858.CD001877.pub2. PMID 17054145
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Agarwal S, Pappas L, Neumayer L, Kokeny K, Agarwal J. Effect of breast conservation therapy vs mastectomy on disease-specific survival for early-stage breast cancer. JAMA Surg. 2014 Mar;149(3):267-74. doi: 10.1001/jamasurg.2013.3049. PMID 24429935
- [Background] Vinh-Hung V, Verschraegen C. Breast-conserving surgery with or without radiotherapy: pooled-analysis for risks of ipsilateral breast tumor recurrence and mortality. J Natl Cancer Inst. 2004 Jan 21;96(2):115-21. doi: 10.1093/jnci/djh013. PMID 14734701
- [Background] Van de Steene J, Soete G, Storme G. Adjuvant radiotherapy for breast cancer significantly improves overall survival: the missing link. Radiother Oncol. 2000 Jun;55(3):263-72. doi: 10.1016/s0167-8140(00)00204-8. PMID 10869741
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155
- [Background] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Background] Veronesi U, Luini A, Del Vecchio M, Greco M, Galimberti V, Merson M, Rilke F, Sacchini V, Saccozzi R, Savio T, et al. Radiotherapy after breast-preserving surgery in women with localized cancer of the breast. N Engl J Med. 1993 Jun 3;328(22):1587-91. doi: 10.1056/NEJM199306033282202. PMID 8387637
- [Background] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Background] Janssen S, Glanzmann C, Lang S, Verlaan S, Streller T, Wisler D, Linsenmeier C, Studer G. Hypofractionated radiotherapy for breast cancer acceleration of the START A treatment regime: intermediate tolerance and efficacy. Radiat Oncol. 2014 Jul 24;9:165. doi: 10.1186/1748-717X-9-165. PMID 25059887
- [Background] Poortmans PM, Collette L, Horiot JC, Van den Bogaert WF, Fourquet A, Kuten A, Noordijk EM, Hoogenraad W, Mirimanoff RO, Pierart M, Van Limbergen E, Bartelink H; EORTC Radiation Oncology and Breast Cancer Groups. Impact of the boost dose of 10 Gy versus 26 Gy in patients with early stage breast cancer after a microscopically incomplete lumpectomy: 10-year results of the randomised EORTC boost trial. Radiother Oncol. 2009 Jan;90(1):80-5. doi: 10.1016/j.radonc.2008.07.011. Epub 2008 Aug 15. PMID 18707785
- [Background] Bartelink H, Maingon P, Poortmans P, Weltens C, Fourquet A, Jager J, Schinagl D, Oei B, Rodenhuis C, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan D, Dubois JB, Remouchamps V, Mirimanoff RO, Collette S, Collette L; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):47-56. doi: 10.1016/S1470-2045(14)71156-8. Epub 2014 Dec 9. PMID 25500422
- [Background] Morgan DA, Robertson JF. Boost or not. J Clin Oncol. 2008 Feb 20;26(6):1013-4; author reply 1014. doi: 10.1200/JCO.2007.15.2017. No abstract available. PMID 18281678
- [Background] https://www.nccn.org/professionals/physician_gls/f_guidelines
- [Result] Fodor A, Brombin C, Mangili P, Borroni F, Pasetti M, Tummineri R, Zerbetto F, Longobardi B, Perna L, Dell'Oca I, Deantoni CL, Deli AM, Chiara A, Broggi S, Castriconi R, Esposito PG, Slim N, Passoni P, Baroni S, Villa SL, Rancoita PMV, Fiorino C, Del Vecchio A, Bianchini G, Gentilini OD, Di Serio MS, Di Muzio NG. Impact of molecular subtype on 1325 early-stage breast cancer patients homogeneously treated with hypofractionated radiotherapy without boost: Should the indications for radiotherapy be more personalized? Breast. 2021 Feb;55:45-54. doi: 10.1016/j.breast.2020.12.004. Epub 2020 Dec 9. PMID 33326894
- [Result] Fodor A, Brombin C, Mangili P, Tummineri R, Pasetti M, Zerbetto F, Longobardi B, Galvan AS, Deantoni CL, Dell'Oca I, Castriconi R, Esposito PG, Deli AM, Rancoita PMV, Fiorino C, Vecchio AD, Di Serio MS, Di Muzio NG. Toxicity of Hypofractionated Whole Breast Radiotherapy Without Boost and Timescale of Late Skin Responses in a Large Cohort of Early-Stage Breast Cancer Patients. Clin Breast Cancer. 2022 Jun;22(4):e480-e487. doi: 10.1016/j.clbc.2021.11.008. Epub 2021 Dec 1. PMID 34955430
- [Result] Bane AL, Whelan TJ, Pond GR, Parpia S, Gohla G, Fyles AW, Pignol JP, Pritchard KI, Chambers S, Levine MN. Tumor factors predictive of response to hypofractionated radiotherapy in a randomized trial following breast conserving therapy. Ann Oncol. 2014 May;25(5):992-8. doi: 10.1093/annonc/mdu090. Epub 2014 Feb 20. PMID 24562444
- [Result] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Result] Coles CE, Haviland JS, Kirby AM, Griffin CL, Sydenham MA, Titley JC, Bhattacharya I, Brunt AM, Chan HYC, Donovan EM, Eaton DJ, Emson M, Hopwood P, Jefford ML, Lightowlers SV, Sawyer EJ, Syndikus I, Tsang YM, Twyman NI, Yarnold JR, Bliss JM; IMPORT Trial Management Group. Dose-escalated simultaneous integrated boost radiotherapy in early breast cancer (IMPORT HIGH): a multicentre, phase 3, non-inferiority, open-label, randomised controlled trial. Lancet. 2023 Jun 24;401(10394):2124-2137. doi: 10.1016/S0140-6736(23)00619-0. Epub 2023 Jun 8. PMID 37302395
- [Result] Pasquier D, Bataille B, Le Tinier F, Bennadji R, Langin H, Escande A, Tresch E, Darloy F, Carlier D, Crop F, Lartigau E. Correlation between toxicity and dosimetric parameters for adjuvant intensity modulated radiation therapy of breast cancer: a prospective study. Sci Rep. 2021 Feb 11;11(1):3626. doi: 10.1038/s41598-021-83159-3. PMID 33574446
- [Result] Brunt AM, Haviland JS, Sydenham M, Agrawal RK, Algurafi H, Alhasso A, Barrett-Lee P, Bliss P, Bloomfield D, Bowen J, Donovan E, Goodman A, Harnett A, Hogg M, Kumar S, Passant H, Quigley M, Sherwin L, Stewart A, Syndikus I, Tremlett J, Tsang Y, Venables K, Wheatley D, Bliss JM, Yarnold JR. Ten-Year Results of FAST: A Randomized Controlled Trial of 5-Fraction Whole-Breast Radiotherapy for Early Breast Cancer. J Clin Oncol. 2020 Oct 1;38(28):3261-3272. doi: 10.1200/JCO.19.02750. Epub 2020 Jul 14. PMID 32663119
- [Result] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Result] Meattini I, Marrazzo L, Saieva C, Desideri I, Scotti V, Simontacchi G, Bonomo P, Greto D, Mangoni M, Scoccianti S, Lucidi S, Paoletti L, Fambrini M, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Pallotta S, Livi L. Accelerated Partial-Breast Irradiation Compared With Whole-Breast Irradiation for Early Breast Cancer: Long-Term Results of the Randomized Phase III APBI-IMRT-Florence Trial. J Clin Oncol. 2020 Dec 10;38(35):4175-4183. doi: 10.1200/JCO.20.00650. Epub 2020 Aug 24. PMID 32840419
- [Result] Coles CE, Aristei C, Bliss J, Boersma L, Brunt AM, Chatterjee S, Hanna G, Jagsi R, Kaidar Person O, Kirby A, Mjaaland I, Meattini I, Luis AM, Marta GN, Offersen B, Poortmans P, Rivera S. International Guidelines on Radiation Therapy for Breast Cancer During the COVID-19 Pandemic. Clin Oncol (R Coll Radiol). 2020 May;32(5):279-281. doi: 10.1016/j.clon.2020.03.006. No abstract available. PMID 32241520